CLINICAL TRIAL: NCT05929989
Title: Role of Cystatin D and Fibrinogen Like Protein 1 in Rheumatoid Arthritis and Their Relation to Disease Activity
Brief Title: Cystatin D Fibrinogen Like Protein 1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba abd el salam selim, dr, Assiut University
Other Study IDs: cystatin D
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Fibrinogen Like Protein 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- active disease
  Interventions: Diagnostic Test: ELISA TEST
- control
  Interventions: Diagnostic Test: ELISA TEST

INTERVENTIONS:
Diagnostic Test: ELISA TEST — ELISA TEST for cystatin D and fibrinogen like protein

SUMMARY:
to detect role of cystatin D and fibrinogen like protein 1 in rheumatoid arthritis asses relationship between disease activity and cystatin D and fibrinogen like protein 1

ELIGIBILITY:
Inclusion Criteria:

* adult patient diagnosed for rheumatoid arthritis

Exclusion Criteria:

* patient with overlap syndrome indiviuals with other auto immune diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patient diagnosed with rheumatoid arthrits
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
detect role of cystatin D and fibrinogen like protein 1 | one year
  detect role of the two biomarkers and there relationship to rheumatoid arthriths

REFERENCES:
- [Background] Lin WW, Ho KW, Su HH, Fang TF, Tzou SC, Chen IJ, Lu YC, Chang MS, Tsai YC, Liu ES, Su YC, Wang YT, Cheng TL, Huang HK. Fibrinogen-Like Protein 1 Serves as an Anti-Inflammatory Agent for Collagen-Induced Arthritis Therapy in Mice. Front Immunol. 2021 Dec 16;12:767868. doi: 10.3389/fimmu.2021.767868. eCollection 2021. PMID 34975855
- [Result] Scherer HU, Haupl T, Burmester GR. The etiology of rheumatoid arthritis. J Autoimmun. 2020 Jun;110:102400. doi: 10.1016/j.jaut.2019.102400. Epub 2020 Jan 22. PMID 31980337